CLINICAL TRIAL: NCT05684094
Title: Mechanisms of Risky Alcohol Use in Young Adults: Linking Sleep Duration and Timing to Reward- and Stress-Related Brain Function
Brief Title: Mechanisms of Risky Alcohol Use in Young Adults: Linking Sleep to Reward- and Stress-Related Brain Function
Acronym: MoRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: University of Pittsburgh (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melynda Casement, Associate Professor of Psychology, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 217901; R01AA029125 (NIH)
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder
Keywords: sleep; circadian; adolescence; substance use; stress; reward
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep extension and advance "Lark Routine" (Experimental): Participants go to bed 90 minutes earlier than their typical average bedtime to extend sleep duration and advance sleep timing
  Interventions: Behavioral: Sleep extension and advance
- Regular sleep duration and timing "Owl Routine" (Active Comparator): Participants go to bed at their typical average bedtime
  Interventions: Behavioral: Regular sleep duration and timing

INTERVENTIONS:
Behavioral: Sleep extension and advance — Participants in the sleep extension and advance condition will maintain a stable sleep schedule that extends sleep duration and advances bedtime by 90 min relative to weekday bedtime. This chronotherapeutic manipulation will include blocking phase-delaying light in the evening using goggles with orange lenses ("blue blockers") beginning 2 h prior to bedtime, and 30 min of 506 lux blue-green light exposure in the morning beginning at rise time using bright light goggles (ReTimer Pty Ltd., Australia). Schedule and chronotherapy adherence will be reinforced using motivational techniques (e.g., securing motivation, preplanning, problem-solving), requiring participants to text the study coordinator and complete morning assessments at rise time, and monetary incentives.
  Arms: Sleep extension and advance "Lark Routine"
Behavioral: Regular sleep duration and timing — Participants in the regular sleep duration and timing condition will keep a stable sleep schedule that matches their typical weekday sleep opportunity and timing. Schedule adherence will be reinforced using motivational techniques (e.g., securing motivation, preplanning, problem-solving), requiring participants to text the study coordinator and complete morning assessments at rise time, and monetary incentives.
  Arms: Regular sleep duration and timing "Owl Routine"

SUMMARY:
This research will use biobehavioral approaches to generate understanding about the linkages between stressful life events, sleep duration and timing, and alcohol use in young adults, with a long-term aim of developing effective preventative interventions for alcohol use disorders.

DETAILED DESCRIPTION:
High-risk drinking (consuming ≥ 4 drinks/day or ≥ 8/week for women, ≥ 5 drinks/day or ≥ 15/week for men) is reported by one in four young adults within the past month and predicts the development and progression of alcohol use disorder (AUD). High-risk drinking can also have terrible costs beyond developing AUD, including death and disability from unintended injuries and suicide attempts, physical and sexual assault, and a wide range of acute and chronic health problems. The high degree of morbidity and mortality associated with high- risk drinking in young adulthood makes this a key developmental period for AUD research and intervention.

High-risk drinking in young adults is related to high exposure to stressors, insufficient sleep duration, and late sleep timing. Alarmingly, almost half of young adults report at least moderate exposure to stressors, only 30% regularly obtain the recommended hours of sleep, and sleep timing is at its latest around age 20. Stressors and short/late sleep may also cause disruptions in reward- and stress-related brain function (e.g., medial prefrontal cortex response to monetary reward, autonomic and neuroendocrine function during stressors), which are key biobehavioral mechanisms of AUD. Short and late sleep habits are a prime target for AUD prevention in young adults; however, there is insufficient causal evidence that improving sleep opportunity and/or timing will alter the biobehavioral mechanisms of AUD or decrease high-risk drinking, particularly in at-risk young adults.

The overall objective of this R01 is to evaluate a biobehavioral model whereby sufficient sleep duration and/or early sleep timing can reduce high-risk drinking by promoting reward- and stress-related brain function in young adults with high lifetime stress load. The long-term goal of this research is to leverage sleep and circadian function to promote mental health. A series of studies by the PI and Co-I Hasler demonstrate that stressful life events, short sleep, and late sleep independently predict future reward- and stress-related brain function and alcohol use and dependence symptoms in adolescents and young adults. However, these studies do not evaluate the additive and interactive effects of stressful life events and sleep/circadian function and do not include experimental designs. More recent research by the PI and Co-I Hasler uses sleep and circadian manipulation to target reward- and stress-related brain function and improve mental health in adolescents and young adults. Building from this research, this R01 will test the central hypothesis that extending and advancing sleep will alter reward- and stress-related brain function in young adults with a history of high-risk drinking and elevated lifetime exposure to stressors. This proposal is consistent with the National Institute on Alcohol Abuse and Alcoholism (NIAAA) Strategic Objective to identify mechanisms underlying AUD and comorbid disorders.

ELIGIBILITY:
Inclusion Criteria:

1. 18-24 years of age;
2. NIAAA criteria for past-month high-risk drinking (i.e., ≥ 4 drinks/day or ≥ 8/week for women, ≥ 5 drinks/day or ≥ 15/week for men);
3. short and late sleep (weekday sleep duration ≤ 7.5 hours and bedtime ≥ 24:00 (midnight); n=60) or long and early sleep (weekday sleep duration > 7.5 hours and bedtime ≤ 24:00 (midnight); n=30);
4. at least moderate lifetime exposure to stressors (≥ 2 events on the 20-item Adult Stress and Adversity Inventory-Screener);
5. not currently in high school; and
6. English language fluency.

Exclusion Criteria:

1. Severe alcohol use disorder (AUD) and/or substance use disorder (SUD), defined as ≥6 AUD/SUD criteria in the Diagnostic and Statistical Manual-5;
2. acute alcohol intoxication on the days of the laboratory post-intensive visits, operationalized as a blood alcohol concentration of .02 or higher during Breathalyzer saliva screen;
3. current clinician-provided diagnosis of narcolepsy or idiopathic hypersomnia;
4. lifetime diagnosis of bipolar or schizophrenia spectrum disorder;
5. certain medical conditions (e.g., serious neurological disorder, heart failure or serious trouble, history of head injury with unconsciousness > 5 minutes);
6. conditions that are contraindicated for MRI (e.g., ferrous metal in the body);
7. positive screen for participant-reported eye disease, epilepsy, or photosensitizing medications that are contraindicated during the manipulation condition when bright light is administered (e.g., psychiatric neuroleptic drugs [e.g., phenothiazine], psoralen drugs, antiarrhythmic drugs [e.g., amiodarone], antimalarial and antirheumatic drugs, porphyrin drugs used in photodynamic treatment of skin diseases);
8. use of melatonin if participant is not willing to discontinue use for the duration of the study.

We will schedule around (i.e., delay appointments as needed) to avoid the timeframe of the following events:

1. urgent suicide risk, defined by moderate/severe risk per CSSR and clinician determination that current risk requires immediate action;
2. travel across two or more time zones within the month prior to the overnight study visits.
3. begin/end a prescribed medication within 2 months of the observational study;
4. medication dose changes within the timeframe calculated as 5x the drug's half-life [the time to reach pharmacokinetic steady-state] before the initiation of the observational or experimental studies;
5. participant-anticipated changes in prescribed medications or medication dosing during the observational or experimental studies.;
6. current symptoms of an airborne infectious illness (e.g., COVID) prior to laboratory visits.

Participants with positive breathalyzer screen (blood alcohol level > .02) will be rescheduled for an alternative overnight visit date.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | 2 months
  The Alcohol Timeline Follow-Back (TLFB) will be administered electronically to assess the quantity (number of standard drinks) and frequency of alcohol use over the past 2 months, beginning at screening and continuing at least every 2 months through the follow-up assessment. The TLFB uses a calendar, anchor dates, and standard drink conversions to obtain retrospective estimates of alcohol use.
Reward-related brain function | 2 weeks
  Functional magnetic resonance imaging (fMRI) during the Monetary Incentive Delay task (MID, 92) will be used to measure blood oxygen level dependent (BOLD) regional response and functional connectivity related to anticipation and receipt of monetary rewards. This task reliably elicits activation in neural reward circuitry
Stress-related brain function | 2 weeks
  Stress-related brain function will be indexed using autonomic and neuroendocrine measures taken before and during the Trier Social Stress Task (TSST). The TSST is a lab-based social-evaluative threat task that reliably elicits subjective stress and increases in the stress-hormone cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Melynda D Casement, PhD, Principal Investigator — University of Oregon
Locations (1):
- Oregon Sleep Lab, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Raw data and data from descriptive/raw measures, as described in the data sharing agreement, will be submitted on a semi-annual basis by July 15 and January 15 or the next business day, beginning on January 15, 2023.
Time Frame: We agree to release and share data in a timely manner, but no later than one year following completion of the funded project period or the date of publication of the main findings from our final data set.
Access Criteria: In order to gain access to data, researchers who were not part of the original research protocol as defined by the University of Oregon Institutional Review Board (IRB) application must submit a detailed description of their project to the Investigator Committee. The proposal must include the investigator's personal identification and institutional affiliation, a current curriculum vita, qualifications, estimated duration of the proposed research, source of financial support, and a conflict of interest statement. The protocol described must include study aims, background and significance, and methods and types of analysis, and a description of the data requested and list of variables. Once approved, the investigator must complete the necessary IRB exempt research application form and document completion of a responsible conduct of research program. Data will not be provided that could identify individual research participants or that the original consent form expressly forbade.